CLINICAL TRIAL: NCT01368003
Title: A Biomarker Study of STA9090 in Castration-Resistant Prostate Cancer (CRPC) With Assessment of Androgen Receptor Pathway Signaling
Brief Title: STA-9090 in Castration-Resistant Prostate Cancer With Assessment of Androgen Receptor Pathway Signaling
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding.
Sponsor: Toni Choueiri, MD (Other)
Responsible Party: Sponsor-Investigator, Toni Choueiri, MD, Overall Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-333
Record Dates: First submitted 2011-04-21; First posted 2011-06-07 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: Castration resistant prostate cancer
MeSH Terms: interventions — STA 9090; Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STA9090 with Dutasteride (Experimental): STA9090 with Dutasteride
  Interventions: Drug: STA9090 with Dutasteride
- STA9090 (Experimental): STA9090
  Interventions: Drug: STA9090

INTERVENTIONS:
Drug: STA9090 — 200 mg/m^2 IV every week for 3 weeks on, 1 week off (days 1,8,15 on a 28-day cycle)
  Arms: STA9090
Drug: STA9090 with Dutasteride — Dutasteride 3.5 mg orally per day STA9090 200 mg/m^2 IV every week for 3 weeks on, 1 week off (days 1,8,15 on a 28-day cycle)
  Other Names: Avodart
  Arms: STA9090 with Dutasteride

SUMMARY:
In this research study, the investigators are looking to determine the safety and efficacy of an investigational drug, STA9090 alone and in combination with dutasteride for the treatment of castrate resistant prostate cancer. STA9090 may cause the growth of cancer to slow down or shrink by targeting proteins required for the cancer to grow. The investigators are also looking to determine whether the use of dutasteride to lower male hormone levels will enhance the effect of STA9090 in the treatment of castrate resistant prostate cancer.

DETAILED DESCRIPTION:
Subjects will have a tumor biopsy before treatment begins. Subjects who are randomized to Arm A will receive infusions of STA9090 on days 1, 8, and 15 of a 28 day cycle. Subjects randomized on Arm B will receive daily oral dutasteride for 2 weeks prior to beginning STA9090 treatment. They will continue to receive dutasteride while on study.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate
* Progressive castration resistant disease
* Metastatic disease
* Normal organ and marrow function

Exclusion Criteria:

* History of current coronary artery disease, myocardial infarction, angina pectoris, angioplasty or coronary bypass
* Current treatment with the following antiarrhythmic drugs: flecainide, moricizine or propafenone
* New York Heart Association class II/III/IV congestive heart failure
* Current or prior radiation therapy to the left hemithorax
* Treatment with chronic immunosuppressants
* Uncontrolled intercurrent illness
* Poor venous access for study drug administration
* Venous thromboembolism in the past 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To assess AR transcriptional activity based on expression of a series of AR regulated genes, in baseline and on therapy tumor biopsies in CRPC patients treated with STA- 9090 +/-dutasteride. | 2 years
  The primary objective is to determine whether STA-9090, or the combination with dutasteride further suppresses AR transcriptional activity. AR transcriptional activity will be assessed based on expression of a series of AR regulated genes, in baseline and on therapy tumor biopsies in CRPC patients treated with STA-9090 +/- dutasteride.

SECONDARY OUTCOMES:
To assess the safety and tolerability of STA9090 in men the CRPC | 2 years
  Each type of toxicity rate (a proportion) will be analyzed and summarized descriptively.
To evaluate progression-free survival (PFS) of men with CRPC treated with STA9090 with or without dutasteride | 2 years
  PFS will be summarized using K-M method.
To evaluate the overall survival of men with metastatic CRPC treated with STA9090 alone or in combination with dutasteride | 2 years
  OS will be summarized using K-M method.
To determine the response rate of measurable disease if present (RECIST) | 2 years
  Patients with measurable disease will be evaluated for response using RECIST criteria and summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Toni K Choueiri, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts